CLINICAL TRIAL: NCT01012843
Title: Does Adjuvant Antibiotic Treatment After Drainage of Anorectal Abscess Prevent the Development of Anal Fistulae? A Prospective Randomized, Placebo Controlled, Double Blind, Multi-Center Clinical Study
Brief Title: Do Antibiotics Prevent Anal Fistulae Formation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Dr. Ulas Sozener, Ankara University School of Medicine Department of General Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AUTF-001
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Anal Fistula
Keywords: Perianal; Abscess; Fistulae in ano; Antibiotic; Anorectal
MeSH Terms: conditions — Rectal Fistula; Abscess | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic (Active Comparator): Patients who received antibiotic treatment after abscess drainage
  Interventions: Drug: Amoxicillin-Clavulanate
- Placebo (Placebo Comparator): Patients who received placebo after abscess drainage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate — oral 875/125 mg tablets of Amoxicillin/Clavulanate 2 times a day for 10 days
  Other Names: Bioment 1 gr BID tablets
  Arms: Antibiotic
Drug: Placebo — oral Placebo tablets two times a day for 10 days
  Arms: Placebo

SUMMARY:
Purpose: This randomized study assesses the effects of antibiotics on the formation of fistulae after drainage of anorectal abscesses.

Methods: Patients who underwent abscess drainage in 3 major colorectal units between September 2005 and January 2008 were included. Previous anorectal surgery history, immunecompromised states, pregnancy, inflammatory bowel disease, antibiotic usage prior to surgery and the presence of an anal fistulae at the time of surgery were the exclusion criteria. Patients were randomized and given either placebo or amoxicillin-clavulanic acid combination treatment for 10 days. Patients were followed one year for perianal fistulae formation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anorectal abscess

Exclusion Criteria:

* Allergy to penicillin derivatives
* Treatment with any antimicrobial agent in the week before enrolment
* Recognized other infection at the time of surgery
* Previous anorectal surgery
* Presence of inflammatory bowel disease
* Suspicion of Fournier's gangrene
* Secondary and recurrent anorectal abscesses
* Presence of an internal opening
* Any additional surgical procedure performed in the same session or during follow-up
* Antibiotic prophylaxis indicated for another reason
* Immunosuppressive and/or anticoagulant drug treatment being taken at the time of surgery
* Diabetes mellitus
* Known chronic disabling disease
* Pregnancy
* Lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Fistula formation | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulas Sozener, M.D., Study Chair — Ankara University
Locations (3):
- Turkey (Türkiye) (3):
  - Ankara Numune Teaching and Research Hospital, Ankara
  - Ankara University School of Medicine Department Of General Surgery, Ankara
  - Dicle University School of Medicine, Diyarbakır

REFERENCES:
- [Background] Vasilevsky CA, Gordon PH. The incidence of recurrent abscesses or fistula-in-ano following anorectal suppuration. Dis Colon Rectum. 1984 Feb;27(2):126-30. doi: 10.1007/BF02553995. PMID 6697831
- [Result] Nunoo-Mensah JW, Balasubramaniam S, Wasserberg N, Artinyan A, Gonzalez-Ruiz C, Kaiser AM, Beart RW Jr, Vukasin P. Fistula-in-ano: do antibiotics make a difference? Int J Colorectal Dis. 2006 Jul;21(5):441-3. doi: 10.1007/s00384-005-0022-4. Epub 2005 Aug 10. PMID 16091913
- [Result] Hamalainen KP, Sainio AP. Incidence of fistulas after drainage of acute anorectal abscesses. Dis Colon Rectum. 1998 Nov;41(11):1357-61; discussion 1361-2. doi: 10.1007/BF02237048. PMID 9823799
- [Result] Ramanujam PS, Prasad ML, Abcarian H, Tan AB. Perianal abscesses and fistulas. A study of 1023 patients. Dis Colon Rectum. 1984 Sep;27(9):593-7. doi: 10.1007/BF02553848. PMID 6468199